CLINICAL TRIAL: NCT05540678
Title: The FibreGum Study - Changing the Course of Obesity in Children
Acronym: FibreGum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: DCB Research AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FibreGum
Record Dates: First submitted 2022-09-05; First posted 2022-09-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nutritional and Metabolic Diseases; Child Obesity; Adolescent Obesity
Keywords: Obesity; Chewing gum; Galactooligosaccharides; GOS (Galactooligosaccharides)
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Chewing gum containing maltitol powder
  Interventions: Dietary Supplement: Placebo
- Investigational (Experimental): chewing gums containing fibers
  Interventions: Dietary Supplement: FibreGum
- No-treatment control (No Intervention): No study chewing gum

INTERVENTIONS:
Dietary Supplement: FibreGum — To chew every day during a period of 6 months 3 chewing gums (morning, noon and evening) for at least 20 minutes each.
  Arms: Investigational
Dietary Supplement: Placebo — To chew every day during a period of 6 months 3 chewing gums (morning, noon and evening) for at least 20 minutes each.
  Arms: Placebo

SUMMARY:
The aim of this study is thus to assess the effect of a chewing gum containing fibres on body weight, metabolism and the oral and intestinal microbiomes in a population of obese children.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent according to International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (ICH/GCP) regulations prior to any study specific procedures
* Obesity as determined by a BMI ≥97th percentile using the Swiss paediatric, age- and sex-matched growth charts
* Newly referred within the last month to a tertiary weight management clinic
* Participant willing to use the study specific monitoring app on his/her own or legal representatives' smartphone

Exclusion Criteria:

* Antibiotic administration in the last 6 months
* Pre- or probiotic treatment in the last 6 weeks
* Any professionally supervised treatment for weight management within the last year
* Consumption of more than one nicotine product per month (e.g. cigarette, gum)
* Adolescent females: any stages of known pregnancy or lactation period
* Congenital disorder affecting the cardiovascular, hepatic or respiratory system in a relevant way (as per PI's or specialist's evaluation)
* Malignant disease on treatment or previous tumour affecting the appetite system (e.g., suprasellar, hypothalamic tumours)
* Systemic antibiotic or anti-inflammatory medication (e.g. systemic intake of glucocorticoids) over the last 7 days
* Known eating disorder (medically diagnosed)
* Participation in another investigation with an investigational drug within the 30 days preceding and during the present investigation
* Dependency from the sponsor or the clinical investigator
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, etc. of the participant and/or legal representative

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in the Body Mass Index (BMI) Z-score | 6 months
  Difference in the BMI Z-scores measured at study start and study completion

SECONDARY OUTCOMES:
Fasting blood glucose change | 6 months
  Differences in fasting blood glucose (mg/dL or mmol/L) between study completion and study start.
Fasting insulin change | 6 months
  Differences in fasting insulin (mIU/mL) between study completion and study start.
HOmeostatic Model Assessment of Insulin Resistance (HOMA-IR) index change | 6 months
  Differences in Homeostatic Model Assessment of Insulin Resistance Index (min:0 - max:10) between study completion and study start. Lower scores mean better outcome.
Hemoglobin A1c (HbA1c) change | 6 months
  Differences in HbA1c (mmol/mol) between study completion and study start.
Lipid-profiles change | 6 months
  Differences in lipid-profiles (Cholesterol, Triglyceride, HDL, LDL in mg/dL) between study completion and study start.
Systolic and diastolic blood pressures changes | 6 months
  Differences in both systolic blood pressure and diastolic blood pressure (mm Hg) between study completion and study start.
Differential blood count change | 6 months
  Differences differential blood count (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils in %) between study completion and study start.
Calprotectin and lipocalin-2 change in stool | 6 months
  Differences in calprotectin and lipocalin-2 (µg/g) in stool between study completion and study start as determined by Enzyme-Linked Immunosorbent Assay (ELISA)
Oral health | 6 months
  Changes in oral microbiota as assessed by 16S ribosomal ribonucleic acid (rRNA) gene sequencing from oral washes.
  Remark: The "S" in 16S is a sedimentation coefficient, that is, an index reflecting the downward velocity of the macromolecule in the centrifugal field.
Intestinal health | 6 months
  Changes in intestinal microbiota-composition as assessed by metagenome sequencing from stool samples
Descriptive analysis of treatment adherence using data from an adherence-tracking app | 6 months
  The assessment of adherence to chewing-gum will be assessed as percentage (%) of chewing-gums chewed.
Alanine Aminotransferase (ALAT) change | 6 months
  Differences in ALAT between study completion and study start.
Calcifediol (25OH-Vitamin D3) change | 6 months
  Differences in Calcifediol between study completion and study start.
Thyroid-Stimulating Hormone (TSH) change | 6 months
  Differences in TSH between study completion and study start.
Ferritin change | 6 months
  Differences in ferritin between study completion and study start.
Proteinuria | 6 months
  Differences in proteinuria between study completion and study start.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Balmer, Prof. med., Study Director — Department of Biomedical Research, Children Clinic Berne, Inselspital, Bern University Hospital University of Bern
Locations (2):
- Switzerland (2):
  - Kinderklinik Bern, Bern
  - Ostschweizer Kinderspital, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No